CLINICAL TRIAL: NCT05603936
Title: Adaption and Testing of the Quality of Life in Short Stature Youth (QoLISSY) Questionnaire for Parents With Children From 0-4
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Bundesverband Kleinwüchsige Menschen und ihre Familien e.V. (Unknown); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: QoLISSY 0-4
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Achondroplasia; Small for Gestational Age; Growth Hormone Deficiency
Keywords: Health related quality of life
MeSH Terms: conditions — Achondroplasia; Dwarfism, Pituitary | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — The original QOLISSY questionnaire was first developed in 2011, it is available as a patient reported and a parent reported instrument. It includes:
  * QoLISSY questionnaire for children and adolescents (8-12, 13-18 yrs)
  * QoLISSY questionnaire for parents of children with short stature (4-7, 8-12 and 13-18 yrs) The QoLISSY instrument can be used to assess the health-related quality of life in short stature youth regardless of its cause; however it was specifically developed for patients with GHD and ISS and their parents.The aim of the current study is the adaption, implementation and validation of the instrument for the investigation of the short stature specific quality of life (QoLISSY) for children (age 0-4 years) with achondroplasia (ACH), Small for Gestational Age (SGA) and Growth Hormone Deficiency (GHD) from a parental perspective.

SUMMARY:
The aim of the study is the adaption, implementation and validation of the instrument for the investigation of the short stature specific quality of life (QoLISSY) for children (age 0-4 years) with achondroplasia (ACH), Small for Gestational Age (SGA) and Growth Hormone Deficiency (GHD) from a parental perspective.

DETAILED DESCRIPTION:
The questionnaire is intended to be particularly applicable in clinical trials, with a focus on the impact of short stature and the physical functionality of those affected. The instrument will be further developed according to the "Guidelines for PRO instrument development". It should be practical in its application and interpretation and applicable in the international context.

In addition, it will be investigated whether, from the parents' point of view, other instruments are suitable for measuring the quality of life of their short statured children. Their preference regarding the instruments will be assessed so that a recommendation can be made as to which instruments are particularly suitable.

A systematic literature review will be conducted to identify suitable instruments to measure the quality of life of short statured children aged 0 to 4.

Approximately 10-20 parents of 0-4 year old children with ACH, GHD and SGA will be recruited for the qualitative data collection (n = 30 to 60). The patients will be recruited through the BKMF (German Association for People of Short Stature and their Families).

In order to test the psychometric properties of the instruments, approximately 30 parents (15 mothers / 15 fathers) of 0-4 year old children with ACH, GHD and SGA will be recruited for the quantitative part of the study (n = 90). All participants will be asked to complete the QoLISSY or other instruments found suitable in the pilot test. For the purpose of cross-validation, the PEDSQL will be used in parallel.

Two weeks after receiving the field test, the re-test will be sent to ensure the reliability of the study. The re-test will be administered to a minimum of 20% of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children aged 0-4 with the diagnosis Achondroplaisa, Short for Gestational Age or Growth Hormone Defiency

Exclusion Criteria:

* Other diagnosis than Achondroplaisa, Short for Gestational Age or Growth Hormone Defiency
* Children older than 4 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents of children aged 0-4 with the diagnosis Achondroplaisa, Short for Gestational Age or Growth Hormone Defiency
Sampling Method: Non-Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life measured by the adapted version of the QoLISSY questionnaire | June 2022 - March 2023
  The studies aim is to identify factors influencing the health related quality of life of children with Achondroplaise, Growth Hormone Deficiency and Small for Gestational Age to adapt and test the QOLISSY-Questionnaire for children from the age of 0-4.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Quitmann, Principal Investigator — Center for Psychosocial Medicine
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No